CLINICAL TRIAL: NCT05771506
Title: Determinants of Balance in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Collaborators: Atlas University (Other)
Responsible Party: Principal Investigator, Hikmet Ucgun, Assistant Professor, Biruni University
Other Study IDs: buhucgun01
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Respiratory Physiological Phenomena; Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD Group: Balance assessment, Pulmonary function test, Respiratory muscle strength test, Peripheral muscle strength test, 6-minute walk test, Cognitive assessment
  Interventions: Other: Balance Assessment; Other: Pulmonary function test; Other: Respiratory muscle strength test; Other: Peripheral muscle strength test; Other: 6-minute walk test; Other: Cognitive assessment
- Control Group: Balance assessment, Pulmonary function test, Respiratory muscle strength test, Peripheral muscle strength test, 6-minute walk test, Cognitive assessment
  Interventions: Other: Balance Assessment; Other: Pulmonary function test; Other: Respiratory muscle strength test; Other: Peripheral muscle strength test; Other: 6-minute walk test; Other: Cognitive assessment

INTERVENTIONS:
Other: Balance Assessment — Balance assessment will be done with the "Biodex Balance System®" (Biodex Medical Systems, Shirley, New York, United States). Postural stability test overall score, stability limits test overall score, and sensory integration test of balance composite score will be recorded.
Other: Pulmonary function test — Pulmonary function test will be performed with a spirometer ("COSMED Pony FX" (COSMED; Italy) in accordance with ATS/ERS criteria. Forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), FEV1/FVC, peak expiratory volume measured at 25% and 75% of forced expiratory time (FEF 25-75%), and peak expiratory volume (PEF) parameters will be measured. The results will be recorded both as a percentage of measured values and expected values.
Other: Respiratory muscle strength test — Respiratory muscle strength will be measured in accordance with ATS/ERS criteria using an electronic, mobile, (MicroRPM, Micro Medical; UK) intraoral pressure measuring device. Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) values will be recorded. Three measurements will be repeated for each maneuver and the highest value recorded as cmH2O.
Other: Peripheral muscle strength test — Peripheral muscle strength will be assessed by measuring M. Quadriceps muscle strength with a digital handheld dynamometer (MicroFET® Hoggan Scientific; USA). The test will be done in three measurements for the dominant side lower extremity. The average of the obtained values will be recorded in kilograms.
Other: 6-minute walk test — Functional capacity will be assessed with the 6-minute walk test (6MWT). 6MWT will be performed in accordance with the criteria of the American Thoracic Society. The 6MWT distance will be recorded in meters.
Other: Cognitive assessment — Cognitive function will be assessed with the Montreal Cognitive Assessment (MoCA) test. The MoCA test is a questionnaire developed to evaluate different cognitive functions and mild cognitive impairment. The maximum score that an individual can obtain from the test is 30, and a score of 21 or above is considered as mild cognitive impairment. Test; will be administered by a certified physiotherapist who has received training on practice and scoring directives

SUMMARY:
The primary aim of our study is to examine the relationship between balance and respiratory function, respiratory and peripheral muscle strength, functional capacity, and cognitive function in patients with Chronic Obstructive Pulmonary Disease (COPD). The secondary aim of our study is to compare respiratory function, respiratory and peripheral muscle strength, functional capacity, balance, and cognitive functions of COPD patients and healthy individuals. This study will examine and record the participant's sociodemographic information and medical records. Balance, respiratory function, respiratory and peripheral muscle strength, functional capacity, and cognitive function will be assessed. Since the patients are included in this study, no intervention will be made, no additional tests will be performed, or no changes will be made in the routine treatments of the patients during the study.

ELIGIBILITY:
COPD Group Inclusion Criteria:

* Being diagnosed with COPD in accordance with the GOLD criteria
* Being between the ages of 40-65
* To be able to speak, read, understand, and cooperate in Turkish
* Being a volunteer to participate in the study

COPD Group Exclusion Criteria:

* Having a COPD exacerbation in the last 8 weeks and/or having an unstable clinical condition
* Having a diagnosed vision, hearing, or neurological disease that may affect balance
* Having any other neurological, orthopedic, cardiovascular, thoracic, or metabolic disease or pathological condition that would affect assessments
* Resting saturation below 90% during exercise tests
* Being on long-term oxygen therapy

Control Group Inclusion Criteria:

* Being between the ages of 40-65
* To be able to speak, read, understand, and cooperate in Turkish
* Being a volunteer to participate in the study

Control Group Exclusion Criteria:

* Having a diagnosed vision, hearing, or neurological disease that may affect balance
* Having any other neurological, orthopedic, cardiovascular, thoracic, or metabolic disease or pathological condition that would affect assessments
* Resting saturation below 90% during exercise tests

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with COPD aged between 40-65 years and healthy adults aged between 40-65 years will be included in the study. Informed consent forms for the study prepared for both the COPD group and the control group will be carefully explained and the participants will be included in the study after they have read, understood, and accepted.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Postural stability test: Overall score | 15-20 minutes
Stability limits test: Overall score | 15-20 minutes
Sensory integration test of balance: Composite score | 20-30 minutes
Forced vital capacity (FVC) | 10-15 minutes
Forced expiratory volume in 1 second (FEV1) | 10-15 minutes
FEV1/FVC | 10-15 minutes
Forced expiratory flow 25-75% (FEF25-75) | 10-15 minutes
Peak expiratory flow (PEF) | 10-15 minutes
Maximal inspiratory pressure (MIP) | 15-20 minutes
Maximal expiratory pressure (MEP) | 15-20 minutes
Quadriceps muscle strength | 15-20 minutes
6-minute walk test | 15-20 minutes
MoCA test | 10-15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No